CLINICAL TRIAL: NCT05417425
Title: A Clinical Study Using Omeza Products in Combination With Standard of Care for the Treatment of Diabetic Foot Ulcers
Brief Title: Omeza Products in Combination With Standard of Care for the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Omeza, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OM-CTP-003.1
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot Ulcers
Keywords: Chronic ulcers; Refractory wounds
MeSH Terms: conditions — Diabetic Foot; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Open-label, single arm to evaluate efficacy of 11 weekly treatments with OCM® in patients with chronic, non-healing Diabetic Foot Ulcers. Percent area reduction (PAR) measurements to be taken at week 5 treatment visit and at week 12 end of study (EOS) visit.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omeza combination therapy and SOC with total contact cast (Experimental): Omeza's products were developed to utilize the benefits of essential omega fatty acids to reduce chronic inflammation and disrupt biofilm colonization commonly found in chronic wounds. The Omeza combination treatment under investigation in this study includes two over the counter (OTC) drugs, Omeza® Lidocaine Lavage and Omeza® Skin Protectant, and a 510(K) medical device, Omeza® Collagen Matrix.
  In combination with standard of care and total contact cast, the products will be applied on a weekly basis. There will be a 14-day screening period to assess chronicity from standard of care alone. At that time treatment will be applied weekly for 4 weeks. Further treatment will be at the discretion of the PI to continue for 8 more weeks or until wound closure.
  Interventions: Combination Product: Omeza collagen matrix, Omeza lidocaine lavage, Omeza skin protectant

INTERVENTIONS:
Combination Product: Omeza collagen matrix, Omeza lidocaine lavage, Omeza skin protectant — The three omeza products were designed to be used in combination for the treatment of chronic wounds

SUMMARY:
This study is to evaluate the efficacy of OCM™ used in combination with off-loading devices for the treatment of diabetic foot ulcers.

DETAILED DESCRIPTION:
The study will include three phases: screening phase, treatment phase and healing confirmation. All measurements in the trial are captured by Tissue Analytics.The two week screening phase is to confirm the chronicity of the diabetic foot ulcer (DFU) and the eligibility of subjects. Subjects will be treated with standard of care (SOC) which includes cleaning of the wound, debridement when needed, dressing, and offloading. If the ulcer decreases by 30% in area measurement after 2 weeks of SOC, then the subject does not qualify for the treatment phase. The treatment phase begins with assessment to confirm continued eligibility and if met, subjects are treated weekly with the OCM™ therapy plus continued offloading. At the conclusion of 4 weekly treatments, the ulcer will be assessed by PI for response and evaluation of percent area reduction. Continued therapy through treatment visit 12 is at the PI's discretion where percent area reduction is assessed and recorded.

OCM™ results will be compared to a Control Group of subjects identified and matched retrospectively from the same site, who received the same advanced treatments that the OCM™ treated cohort had received prior to the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old and female subjects are not pregnant
* Subject is diagnosed as having Type 1 or Type 2 diabetes
* Presence of a DFU, Wagner 1 or 2, extending at least through the dermis, provided it is below the level of the medial or lateral malleolus
* Target wound will be located on the foot or ankle and will be the largest ulcer if two or more DFUs are present with the same Wagner grade and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2cm distant from the target wound.
* Study ulcer has been present for at least 1 month and less than or equal to 12 months as of the date the subject signs consent for study
* Study ulcer size is a minimum of 1.0 cm2 and a maximum of 100.0 cm2
* Study ulcer may have characteristics that include yellow/white slough with or without fibrous/scar tissue and/or non-viable tissue, but not mandatory
* Subject understands and is willing to participate in the clinical study including offloading prior to study start, participate in the informed consent process, and can comply with weekly visits and the follow-up regimen
* Willing and able to comply with study procedures, including study visits and study dressing regimens
* Subject has read and signed the IRB-approved Informed Consent Form before screening procedures are undertaken

Exclusion Criteria:

* Study ulcer deemed by the Investigator to be caused by a medical condition other than Diabetes
* Study ulcer exhibits clinical signs and symptoms of infection, as evidenced by tissue necrosis, redness, pain, and/or purulent drainage and/or receiving systemic antibiotics for the treatment of such
* Study ulcer is treated with a topical antibiotic during the screening phase
* Study ulcer requires enzymatic debridement during the study
* Study ulcer is less than 2.0 cm2 or greater than 100.0cm2
* Study ulcer has been treated with tissue engineered material (e.g., Apligraf® or Dermagraft®) or other scaffold materials (e.g., Oasis, PuraPly AM or Matristem) within the last 30 days
* Study ulcer requiring negative pressure wound therapy or hyperbaric oxygen during the course of the trial
* Study ulcer decreases in area by 30% or more during the 14 days screening period
* Presence of any condition(s) that seriously compromises the subject's ability to complete this study.
* Subjects with a BMI>65
* Subject is an active smoker
* Subject has any history of fish allergy or a known sensitivity to any of the SoC materials which come into contact with the skin
* Subject is on Dialysis
* Any active cancer other than a nonmelanoma skin cancer; any previous cancer must be in remission for at least 1 year: bone cancer of metastatic disease of the affected limb, or has had chemotherapy within the last 12 months
* Suspicion of malignancy. If a clinical suspicion of malignancy exists in the opinion of the Investigator, a biopsy should be performed regardless of duration of wound.
* Life expectancy < 6 months
* Subject has received within 28 days of screening a treatment which is known to interfere with or affect the rate and quality of wound healing (e.g., thrombolysis, systemic steroids, immunosuppressive therapy, autoimmune disease therapy, dialysis, radiation therapy, chemotherapy, revascularization surgery) and who may receive such medications during the screening period or who has anticipated to require such medications during the course of the study
* History of immunodeficiency or any illness or condition that could interfere with wound healing e.g., lymphedema, end-stage renal disease, severe malnutrition, liver disease, aplastic anemia. Raynaud's Syndrome, connective tissue disorder, acquired immune deficiency syndrome, connective tissue disorder, acquired immune deficiency syndrome, HIV positive, or sickle cell anemia
* Untreated osteomyelitis or bone infection of the affected foot as verified by x-ray within 30 days prior to treatment. (In the event of an ambiguous diagnosis, the subject will not be enrolled)
* Hepatitis
* Acute deep venous thrombosis
* Allergy to lidocaine and/or epinephrine
* Subject's inability to safely ambulate with the use of the study-required off-loading method
* Subject has unstable Charcot foot or Charcot with bone exposed that could inhibit wound healing
* All females of childbearing potential who are not using a highly effective method of birth control (failure rate less than 1% per year), such as implants, injectables, combined oral contraceptives, some IUDs, practice sexual abstinence or have a vasectomized partner.
* The following are prohibited within 30 days prior to randomized treatment and throughout the study: Heat lamps, UV lights, Whirlpool baths, Hyperbaric oxygen, Jet water streams (other than gentle saline irrigation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Percent area change after 4 weeks of treatment compared to baseline | 6 weeks
  After a 2 week screening phase with standard of care and total contact casting, the wound will be measured and assessed by Tissue Analytics platform. At each treatment visit the change in the wound size and healing status will be assessed. After 4 weeks of treatment the change in wound size will be compared to baseline measurement from treatment visit 1 and the percent area reduction (PAR) recorded.
Incidence in wound closure by week 12 of treatment | 14 weeks
  Treatment will continue and measurements recorded by Tissue Analytics platform until wound closure or up to 12 weeks of treatment.

SECONDARY OUTCOMES:
Incidence of adverse events | 14 weeks
  Safety of the products used in combination will be assessed by the PI and assesses throughout treatment for adverse events or reactions to the products.
Change in subject's perception of pain at baseline and weekly throughout treatment | 14 weeks
  Subjects will be required to assess ulcer pain at baseline and at each treatment visit by a questionnaire assessing pain on a numerical scale
Increase in physical function and ambulation | 14 weeks
  Subjects will be asked to complete a questionnaire to assess physical function and ambulation status at baseline and at each treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Simman, MD, Principal Investigator — ProMedica Physician Group
Locations (1):
- Jobst Vascular Institute, Toledo, Ohio, United States